CLINICAL TRIAL: NCT00288028
Title: A Phase I Study of Bortezomib During Maintenance Phase After High Dose Melphalan and Autologous Stem Cell Transplantation in Patients With Multiple Myeloma
Brief Title: Bortezomib in Treating Patients With Multiple Myeloma Who Have Undergone an Autologous Peripheral Blood Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Muneer Abidi, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000455585; P30CA022453 (NIH); WSU-D-2957; WSU-0506002467
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib (Experimental): Bortezomib is administered as a 5 second IV bolus on days 1, 4, 8,11 or 1,8 and 15 of a 21-35 days cycle (Depending on the Dosing schedule). The dosage will be calculated based on actual weight of the patient unless the actual weight is greater than 40% above the ideal body weight. In this instance the dosage will be based on the adjusted ideal body weight. The Adjusted IBW (kg) = IBW + 0.25 x (actual body weight - IBW). The dosage will be adjusted based on the safety and toxicity profile, until a MTD is determined.
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — Dose of Bortezomib* Level 1: 1.3 mg/m2 on Day 1, 4, 8, 11 - Every 21 days; Level 2: 1.3 mg/m2 on Day 1, 4, 8, 11 - Every 28 days; Level 3: 1.0 mg/m2 on Day 1, 8, 15 - Every 28 days; Level 4: 1.0 mg/m2 on Day 1, 8, 15 - Every 35 days
  Other Names: Velcade®

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving bortezomib after an autologous peripheral blood stem cell transplant may stop the growth of any cancer cells that remain after transplant.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib in treating patients with multiple myeloma who have undergone an autologous peripheral blood stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of bortezomib during maintenance phase after high-dose melphalan and autologous peripheral blood stem cell transplantation in patients with multiple myeloma.
* Determine the safety and tolerability of bortezomib in these patients.

Secondary

* Determine the overall response rate, complete response rate, and response duration in patients treated with bortezomib at the MTD.

OUTLINE: This is an open-label, dose-finding study.

Patients receive bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 21 or 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive de-escalating doses of bortezomib (at varying dosing schedules) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

After completion of study treatment, patients are followed at 1 year.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma
* Must have completed high-dose melphalan and autologous peripheral blood stem cell transplantation

  * Transplant must have been completed 30-120 days ago
  * Must not be receiving maintenance therapy
  * Patients must have received 200 mg/m² of melphalan intravenously as a conditioning regimen (no dose reduction allowed)
* No evidence of amyloidosis
* No available donor

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 or Karnofsky PS 60-100%
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 75,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal
* Transaminase ≤ 3 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must have a negative HIV test
* No baseline neurological disease > grade I
* No cranial nerve palsy
* No demonstrated resistance to bortezomib
* No history of allergic reactions attributed to bortezomib, boron, or mannitol
* No cardiac arrhythmia
* No unstable angina pectoris
* No symptomatic congestive heart failure
* No ongoing or active infection
* No other uncontrolled illness
* No psychiatric illness or social situations that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No other concurrent anticancer therapies or agents
* No other concurrent investigational agents
* Not receiving maintenance therapy after prior stem cell transplantation on another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-07; Primary Completion 2010-11 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | At course 8
Safety and tolerability | At course 8

SECONDARY OUTCOMES:
Overall response rate by Southwest Oncology Group (SWOG) criteria | At day 30 following stem cell transplant and following course 4, course 8, and 1 year of study treatment
Complete response rate by SWOG criteria | At day 30 following stem cell transplant and following course 4, course 8, and 1 year of study treatment
Response duration by SWOG criteria | At day 30 following stem cell transplant and following course 4, course 8, and 1 year of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Muneer H. Abidi, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States